CLINICAL TRIAL: NCT00619255
Title: Maternal Child Health Bureau Adolescent Trauma Recovery and Stress Disorders Collaborative Care (ATRSCC) Model Program Trial
Brief Title: Adolescent Trauma Recovery and Stress Disorders Collaborative Care (ATRSCC) Model Program Trial
Acronym: ATRSCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32685; 1 H34 MC08508-01-00; 07-7850-C01 (Other: University of Washington)
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Post-traumatic Stress Disorder; Alcohol Abuse; Alcohol Dependence
Keywords: Adolescents; Quality Assurance and Improvement; Substance Abuse; Posttraumatic Stress; Family Centered Care; Trauma Systems
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Adolescent Trauma Support Program
  Interventions: Behavioral: Adolescent Trauma Support Program
- Control (No Intervention): Usual Care Control Condition

INTERVENTIONS:
Behavioral: Adolescent Trauma Support Program — The study team will be organized into an adolescent trauma support service. The adolescent trauma support service will fundamentally restructure psychosocial care by integrating post-injury medical treatment with alcohol and PTSD detection and treatment. The adolescent trauma support specialists will deliver a stepped collaborative care intervention to adolescents and their families over the 6-12 months post-injury.
  Arms: Intervention

SUMMARY:
Recent needs assessments suggest that difficulties exist in care coordination between emergency medical services (EMS) systems and primary care for injured adolescents with alcohol problems and post-traumatic stress disorder (PTSD). This project will implement, evaluate, and disseminate the adolescent trauma support service model program that aims to enhance coordination between EMS systems and primary care/community services.

DETAILED DESCRIPTION:
Goal 1: To coordinate care from EMS systems to primary care for injured adolescents.

Objective 1: To increase rates of connection to primary care providers to 55% for model program adolescents, compared to an anticipated connection rate of 25% in adolescents assigned to standard care, by 2010.

Goal 2: To reduce alcohol consumption over the course of the year after injury.

Objective 2: To reduce rates of alcohol consumption by 25% in adolescents assigned to the model program, compared to adolescents assigned to the standard care, by 2010.

Goal 3: To reduce adolescent PTSD symptoms over the course of the year after injury.

Objective 3: To achieve statistically significant reductions in PTSD symptoms in model program patients, compared to adolescents assigned to standard care, by 2010.

Activities Undertaken to Meet Project Goals:

We propose to implement and evaluate an innovative model program, the adolescent trauma support service, that aims to improve the quality of care for injured adolescents with problematic alcohol use and high levels of PTSD symptoms by enhancing coordination of care between EMS systems and primary care and community services. All injured adolescents ages 12-18 presenting to the Harborview Medical Center with injuries so severe that they require inpatient admission and/or 24 hour observation in the emergency department, will be screened for alcohol use and PTSD. Adolescents who screen into the study will be randomly assigned to the adolescent trauma support service or standard care. Two trauma support specialists will meet each injured adolescent and available family members by the ED gurney or inpatient bedside in order to elicit and address each patient/family's unique constellation of post-injury concerns. Next, the adolescent trauma support specialist will help to coordinate care received within the EMS system with primary care providers. The trauma support specialists will also have the capacity to deliver evidence-based motivational interviewing interventions targeting reductions in adolescent alcohol use. The trauma support specialists will link patients and families to evidence-based PTSD treatment through primary care and community resources. Program evaluation will include a comparison of the outcomes of adolescents randomly assigned to the adolescent trauma support program with those of adolescents assigned to standard care. Adolescents in the model program and standard care will be compared on the presence or absence of post-injury primary care visits and reductions in alcohol use and PTSD symptoms over the course of the year after injury. Nationwide dissemination activities of program evaluation results will include the publication of manuscripts in peer reviewed journals and presentations at national meetings by members of the interdisciplinary collaborative group that includes pediatric, mental health and surgical providers.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will screen all English speaking female and male adolescents ages 12-18, who present to Harborview Medical Center with injuries so severe that they require inpatient admission and/or > 24 hour observation in the emergency department.
* All dyads where both parents consent and adolescents assent to the study will be enrolled in the study and randomized.

Exclusion Criteria:

* Adolescents who have suffered head, spinal cord, or other severe injuries that prevent participation in the baseline interview will be excluded from the protocol.
* Patients who require immediate intervention (e.g., self-inflicted injury, active psychosis, mania, and victims of family abuse) will be excluded and referred to the Harborview Inpatient Psychiatric Consult Service.
* Patients who are currently incarcerated or are likely to face criminal charges will be excluded.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2010-10-31 (Actual); Study Completion 2014-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas F. Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Zatzick D, Russo J, Lord SP, Varley C, Wang J, Berliner L, Jurkovich G, Whiteside LK, O'Connor S, Rivara FP. Collaborative care intervention targeting violence risk behaviors, substance use, and posttraumatic stress and depressive symptoms in injured adolescents: a randomized clinical trial. JAMA Pediatr. 2014 Jun;168(6):532-9. doi: 10.1001/jamapediatrics.2013.4784. PMID 24733515
- See also: Our study is no longer recruiting, if you are seeking care for PTSD from Harborview Medical Center please follow this link. — http://depts.washington.edu/hcsats/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 59 | 61
Completed | 57 | 61
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (1.9) | 15.4 (1.9) | 15.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 45 | 45 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 52 | 56 | 108
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 37 | 42 | 79
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With High Levels of Adolescent PTSD Symptoms
Description: Patients with symptoms consistent with a diagnosis of PTSD on the UCLA PTSD Reaction Index were counted. The UCLA PTSD-RI can be used to create an algorithm consistent with a diagnosis of PTSD by rating 1 intrusive, 3 avoidant, and 2 arousal symptoms with a rating of moderate severity. The PTSD-RI is scored on a scale from 0 (none of the time) - 4 (most of the time) with a > = 2 "some of the time" denoting this cutoff for moderate severity. This algorithm was used to identify patients with high PTSD symptom levels consistent with a diagnosis of PTSD.
Time Frame: Baseline (injury), then 2, 5, and 12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 61
Participants
  Baseline | 9 | 12
  2-months | 11 | 12
  5-months | 9 | 13
  12-months | 12 | 9
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.71, Chi-squared; DF=3; Slope = 1.38

2. Secondary Outcome: Number of Patients Who Self-reported Alcohol Consumption or Drug Use
Description: Any self-reported alcohol or drug use using one yes or no question
Time Frame: Baseline (injury), and 2, 5, and 12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 61
Participants
  Baseline | 28 | 25
  2-months | 18 | 14
  5-months | 19 | 21
  12-months | 22 | 26
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.80, Chi-squared; DF=3; Slope = 1.02

3. Secondary Outcome: Percentage of Asolescents Linked to Primary Care During the Study
Description: Percentage of adolescents self-reporting one or more primary care visits over the course of the 12-months after the injury
Time Frame: Up to12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 61
Participants | 43 | 48
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.67, Chi-squared; DF = 1 Chi-Square Value = 0.18

4. Secondary Outcome: Percentage of Adolescents Who Self-reported Weapon Carriage
Description: Self-reported carrying of knife, gun, club or other weapon by adolescent
Time Frame: Baseline (injury), then 2, 5, and 12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 61
Participants
  Baseline | 20 | 19
  2-months | 8 | 15
  5-months | 5 | 13
  12-months | 4 | 13
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.03, Chi-squared; DF=3; Slope = 9.0

5. Secondary Outcome: Number of Patients Experiencing High-Level Depressive Symptoms
Description: The investigators used the Patient Health Questionnaire (PHQ-9) to identify symptoms consistent with a diagnosis of depression on the 9-item Patient Health Questionnaire depression screen. Scores range from 1 to 27 with higher scores representing worse outcomes.
Time Frame: Baseline (injury), then 2, 5, and 12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 61
Participants
  Baseline | 4 | 8
  2-months | 3 | 4
  5-months | 2 | 4
  12-months | 7 | 6
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.72, Chi-squared; DF=3; Slope = 1.35

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 14/59 | 13/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=59) | Control (N=61)
Suicide ideation (Psychiatric disorders) | 14 | 13 — PHQ-9 Score of >0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No